CLINICAL TRIAL: NCT04632329
Title: Negative Pressure Applied by the Equinox Mercury™ Multi-Pressure Dial to Lower and Modulate Intraocular Pressure in Subjects With Severe Open Angle Glaucoma (The Ranger Study)
Brief Title: Negative Pressure Applied by the Equinox MPD for Severe Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Equinox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: CP-022
Record Dates: First submitted 2020-10-31; First posted 2020-11-17 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Negative Pressure (Experimental)
  Interventions: Device: Negative Pressure Treatment via the Mercury Multi-Pressure Dial
- Control Eye (No Intervention)

INTERVENTIONS:
Device: Negative Pressure Treatment via the Mercury Multi-Pressure Dial — Negative Pressure Treatment via the Mercury Multi-Pressure Dial
  Arms: Negative Pressure

SUMMARY:
This is a prospective, non-significant risk, controlled, randomized, multi-center, masked, feasibility study to evaluate the safety and IOP-lowering effectiveness of negative pressure application (via the Mercury MPD) for lowering and titrating intraocular pressure (IOP) in severe open-angle glaucoma (OAG) patients. The study will be conducted at approximately three investigational sites in the United States. Between 60 and 100 subjects will be randomized to treatment. Treatment eyes will be administered two levels of negative pressure, calculated based on 50% and 75% of baseline IOP (as measured by pneumatonometry). One eye of each eligible subject will be randomized to receive negative pressure application with the MPD device; the contralateral eye will be used as a control and will be examined but will not undergo application of negative pressure. Subjects will be treated at each of the negative pressure levels for one hour. All study procedures will be conducted at one visit, and the subject will exit the study at the conclusion of the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 22 years of age at the time of signing the informed consent
2. Subjects willing to sign the informed consent and capable of committing to the study assessments
3. Subjects with orbital anatomy that permits a proper seal in both eyes when goggles are placed over eyes and can obtain IOP measurements with Excursion goggles in place
4. Subjects with a diagnosis of severe open-angle glaucoma (OAG definition is inclusive of primary open angle glaucoma, normal tension glaucoma, pseudoexfoliative glaucoma, and pigmentary glaucoma) in at least one eye, defined by glaucomatous optic disc or RNFL abnormalities AND visual field abnormalities in both hemifields and/or loss within 5 degrees of fixation in at least one hemifield as tested with standard automated perimetry (the diagnosis of the contralateral eye may include suspected OAG< as well as mild/moderate/severe OAG)
5. Subjects with treatment regimens including current ocular hypotensive medications, prior non-incisional surgical procedures (e.g. MIGS and SLT), or any combination of the two
6. Subjects who are literate, able to speak English or Spanish, and able to understand and follow study instructions

Exclusion Criteria:

1. Subjects with a history of allergy to primary study device material (i.e., silicone and latex)
2. Subjects with a history of any ocular disorder or condition (e.g., corneal transplant) in either eye that would likely interfere with the interpretation of the study results or compromise subject safety
3. Subjects with a history of retinal tear/detachment, wet macular degeneration, diabetic macular edema, or proliferative diabetic retinopathy
4. Subjects with active conjunctival chemosis or anterior uveitis
5. Subjects with a Van Herick grade of 2 or less.
6. Subjects with a history of prior incisional filtering (i.e. trabeculectomy) or tube/shunt glaucoma surgery in either eye
7. Subjects with best corrected visual acuity of 20/200 or worse in either eye due to glaucoma
8. Subjects who do not wish to or cannot comply with study procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
IOP* reduction of ≥ 20% with 50% Negative Pressure for the treatment group vs. the control group | Day 1
  Feasibility to lower intraocular pressure inside the eye in 1 treatment session (1-day). Not a measure of glaucoma progression health outcome. Difference in IOP as measured via pneumatonometry with Excursion goggles worn immediately before vs. during application of negative pressure.
Mean IOP*reduction with 50% Negative Pressure for the treatment group vs. the control group | Day 1
  Feasibility to lower intraocular pressure inside the eye in 1 treatment session (1-day). Not a measure of glaucoma progression health outcome. *Difference in IOP as measured via pneumatonometry with Excursion goggles worn immediately before vs. during application of negative pressure

SECONDARY OUTCOMES:
IOP* reduction of ≥ 25% with 75% Negative Pressure for the treatment group vs. the control group | Day 1
  *Difference in IOP as measured via pneumatonometry with Excursion goggles worn immediately before vs. during application of negative pressure
Mean IOP*reduction with 75% Negative Pressure for the treatment group vs. the control group | Day 1
  *Difference in IOP as measured via pneumatonometry with Excursion goggles worn immediately before vs. during application of negative pressure

OTHER OUTCOMES:
Adverse Biomicroscopic Slit Lamp Findings | Day 1
  Slit lamp findings before and after negative pressure applications
Rate of ocular/periocular adverse events (% by adverse event) | Day 1
  Safety Outcomes
Corrected Distance Visual Acuity | Day 1
  Safety Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Nate Radliffe, MD, Study Director — New York Eye Surgery Center
Locations (3):
- United States (3):
  - Illinois College of Optometry, Chicago, Illinois
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - R and R Eye Research, LLC, San Antonio, Texas